CLINICAL TRIAL: NCT00727714
Title: Circulating Inflammatory Markers, Exhaled NO and Lung Function in Cement Production Workers; a Cross-shifts Study
Brief Title: Lung Function and Inflammatory Markers in Cement Dust Exposed Workers: A Cross-shifts Study
Acronym: LIS
Status: Completed | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Rikshospitalet University Hospital (Other); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anne Kristin M. Fell, Senior physician, MD, PhD, Sykehuset Telemark
Other Study IDs: STHF 5690.11, REK S-08083a
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Airway Obstruction
Keywords: Cement dust exposure; Cross-shift study; Lung function indices; Exhaled nitric oxide; Serum inflammatory markers
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to examine possible changes in lung function, nitric oxide levels and systemic inflammatory markers in cement dust exposed workers, during one shift (6-8 hours).

DETAILED DESCRIPTION:
OBJECTIVE:

Cement dust is suspected to be one of the main factors causing increased mortality among workers not only in the cement production industry, but also in the construction industry worldwide. Our aim is to examine possible changes in lung function, nitric oxide levels and systemic inflammatory markers in cement dust exposed workers, during one shift (6-8 hours).

METHODS:

All employees from Norwegian cement plants, are invited to participate. The workers will perform spirometry, single-breath determination of carbon monoxide uptake, blood samples before and after a working shift of 6-8 hours, and again after 24 hours. Information on respiratory symptoms, allergy and former respiratory disease as well as exposure information will be given on a self-reported questionnaire. Changes in lung function indices, nitric oxide levels and serum inflammatory markers will be calculated. Nitric oxide will only be measured in non-smokers. We will compare cement dust exposed workers with low-level or non-exposed workers (controls).

ELIGIBILITY:
Inclusion Criteria:

* Employees from a Norwegian cement production plant

Exclusion Criteria:

* Exhaled nitric oxide measurements: smokers
* Substantial previous work in quarry or as a miner

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All employees of two Norwegian cement production plants are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johny Kongerud, MD, PhD, Study Chair — Rikshospitalet University Hospital; Helge Kjuus, MD, PhD, Study Chair — National Institute of occupational Health, NIOH; Marit Skogstad, MD, PhD, Principal Investigator — National Institute of occupational Health, NIOH
Locations (1):
- Sykehuset Telemark HF, Skien, Norway

IPD SHARING:
Plan to Share IPD: No
The individual data is no longer available, due to regulations in Norway requiering individual data to be deleted 5 years after the study was compleeted.

REFERENCES:
- [Background] Abrons HL, Petersen MR, Sanderson WT, Engelberg AL, Harber P. Symptoms, ventilatory function, and environmental exposures in Portland cement workers. Br J Ind Med. 1988 Jun;45(6):368-75. doi: 10.1136/oem.45.6.368. PMID 3260798
- [Background] Fell AK, Thomassen TR, Kristensen P, Egeland T, Kongerud J. Respiratory symptoms and ventilatory function in workers exposed to portland cement dust. J Occup Environ Med. 2003 Sep;45(9):1008-14. doi: 10.1097/01.jom.0000083036.56116.9d. PMID 14506344
- [Background] Ali BA, Ballal SG, Albar AA, Ahmed HO. Post-shift changes in pulmonary function in a cement factory in eastern Saudi Arabia. Occup Med (Lond). 1998 Nov;48(8):519-22. doi: 10.1093/occmed/48.8.519. PMID 10024727
- [Background] Larsson K. Aspects on pathophysiological mechanisms in COPD. J Intern Med. 2007 Sep;262(3):311-40. doi: 10.1111/j.1365-2796.2007.01837.x. PMID 17697154
- [Background] Raulf-Heimsoth M, Pesch B, Schott K, Kappler M, Preuss R, Marczynski B, Angerer J, Rihs HP, Hahn JU, Merget R, Bruning T. Irritative effects of fumes and aerosols of bitumen on the airways: results of a cross-shift study. Arch Toxicol. 2007 Jan;81(1):35-44. doi: 10.1007/s00204-006-0115-z. Epub 2006 May 19. PMID 16710697
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Macintyre N, Crapo RO, Viegi G, Johnson DC, van der Grinten CP, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, Gustafsson P, Hankinson J, Jensen R, McKay R, Miller MR, Navajas D, Pedersen OF, Pellegrino R, Wanger J. Standardisation of the single-breath determination of carbon monoxide uptake in the lung. Eur Respir J. 2005 Oct;26(4):720-35. doi: 10.1183/09031936.05.00034905. No abstract available. PMID 16204605
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 95 workers from two cement plants in Norway (located in the small cities of in Brevik in South-Norway and Kjøpsvik in the North-Norway) were examined in the winter sesons in 2008 and 2009.
Pre-assignment Details: The workers were required to be off work for at least two days before Medical examinations, then exposed to cement Production dust between 0 and 8 h and again between 24 and 32 h. Those not exposed in these periods were excluded. No unexposed controls were included, the participants were their own controls.
Groups:
- Exposed Workers: 95 workers from two cement plants in Norway were included and examined pre and post shift (ohr and 8hr)and again after 24 hours.
Period: Overall Study
Arm/Group | Exposed Workers
Started | 95
Completed | 93
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Exposed Workers
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 88
Region of Enrollment [Number; unit: participants]
  Norway | 95
height [Mean (Standard Deviation); unit: cm] | 179 (7)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28 (4)
Smoking [Number; unit: participants]
  Never-smokers | 34
  Ex-smokers | 22
  Smokers | 39
duration of exposure [Mean (Standard Deviation); unit: years] | 16 (13)
Spirometry [Mean (Standard Deviation); unit: Litres]
  FVC | 5.02 (0.91)
  FEV1 | 3.92 (0.81)
Fraction of exhaled nitric oxide (FeNO) [Median (Full Range); unit: parts per billion] | 14 [0 to 96]
Inflammatory markers in blood [Median (Full Range); unit: ng/litre]
  IL-1B | 0.25 [0.09 to 7.00]
  IL-10 | 1.12 [0.18 to 10.78]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Lung Function Measurements During One Work Shift (6-8h)
Description: Changes in lung function measurements during one work shift (6-8h), spirometry and gass diffusion capacity
Time Frame: baseline and 6-8h
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Exposed Workers
Number analyzed (Participants) | 93
Litres
  FVC | 4.99 (0.97)
  FEV1 | 3.88 (0.81)

2. Secondary Outcome: Changes in FeNO Measurements During One Shift (6-8h)
Time Frame: baseline and 6-8h
Population: Problems With the FeNO (NIOX) device lead to few (58) included in FeNO measurements
Measure: Median (Full Range); unit: ppb
Arm/Group | Exposed Workers
Number analyzed (Participants) | 58
ppb | 14 [0 to 98]

3. Secondary Outcome: Changes in Serum/Plasma Inflammatory Markers During One Shift (6-8h)
Time Frame: Baseline and 6-8h
Measure: Median (Full Range); unit: ng/Litre
Arm/Group | Exposed Workers
Number analyzed (Participants) | 88
ng/Litre
  IL-1B | 0.23 [0.09 to 3.51]
  IL-10 | 0.91 [0.09 to 6.45]

4. Secondary Outcome: Changes in FeNO Measurements Between Baseline (0h) and 32 h
Time Frame: 0-32h
Measure: Median (Full Range); unit: ppb
Arm/Group | Exposed Workers
Number analyzed (Participants) | 58
ppb | 12 [0 to 82]

5. Secondary Outcome: Changes in Serum/Plasma Inflammatory Markers Between Baseline and 32 h
Time Frame: 0-32h
Measure: Median (Full Range); unit: ng/Litre
Arm/Group | Exposed Workers
Number analyzed (Participants) | 88
ng/Litre
  IL-1B | 0.20 [0.09 to 3.51]
  IL-10 | 0.97 [0.10 to 4.55]

ADVERSE EVENTS:
Time Frame: Two weeks
Arm/Group | Exposed Workers
Serious Adverse Events (participants affected / at risk) | 0/95
Other Adverse Events (participants affected / at risk) | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes